CLINICAL TRIAL: NCT05486572
Title: CSP #2023 - Preventing Liver Cancer Mortality Through Imaging With Ultrasound vs. MRI (The PREMIUM Study)
Brief Title: Preventing Liver Cancer Mortality Through Imaging With Ultrasound vs. MRI
Acronym: PREMIUM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Carcinoma, Hepatocellular; Cirrhosis
Keywords: hepatic, oncology; liver; chronic diseases; health services and systems; prospective, randomized, clinical trial; magnetic resonance imaging; ultrasonography; cirrhosis; liver cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Fibrosis; Neoplasms; Chronic Disease; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abdominal Ultrasound Screening with serum AFP (Active Comparator): abdominal ultrasound (US)+serum alpha fetoprotein (AFP) every 6 months from the time of recruitment until the end of year 8
  Interventions: Other: Abdominal Ultrasound Screening with serum AFP
- Abbreviated Magnetic Resonance Imaging with serum AFP (Other): Abdominal aMRI+ serum AFP every 6 months from the time of recruitment until the end of year 8
  Interventions: Other: Abbreviated Magnetic Resonance Imaging with serum AFP

INTERVENTIONS:
Other: Abbreviated Magnetic Resonance Imaging with serum AFP — Abdominal aMRI+ serum AFP every 6 months from the time of recruitment until the end of year 8
  Arms: Abbreviated Magnetic Resonance Imaging with serum AFP
Other: Abdominal Ultrasound Screening with serum AFP — abdominal ultrasound (US)+serum alpha fetoprotein (AFP) every 6 months from the time of recruitment until the end of year 8
  Arms: Abdominal Ultrasound Screening with serum AFP

SUMMARY:
The study is a randomized trial of two different screening methods for early detection of liver cancer in patients with cirrhosis of the liver. The goal of PREMIUM is to compare an abbreviated version of the diagnostic gold standard for HCC (aMRI) +AFP to the standard-of-care screening (US+AFP) in patients at high risk of developing HCC. The investigators hypothesize that HCC will be detected at earlier stages, allowing for more curative treatments and resulting in a reduction in HCC-related mortality.

DETAILED DESCRIPTION:
Study Design. The investigators propose to conduct a randomized controlled trial of screening for hepatocellular carcinoma (HCC) by ultrasound (US)+serum alpha fetoprotein (AFP) every 6 months (the current standard-of-care) versus abbreviated MRI (aMRI)+AFP every 6 months among patients with cirrhosis who have a high risk of HCC (estimated annual HCC risk >2.5%).

Study Population. Patients ages 18-75 with cirrhosis (standard histologic, radiologic, or clinical criteria) of any etiology, with estimated annual HCC risk >2.5%. Exclusion Criteria: Prior HCC; Child C Cirrhosis (CTP score 10); MELD score >20; Listed for liver transplantation; Contra-indications to MRI; Comorbidities with limited life expectancy defined by a cirrhosis-specific comorbidity index (CirCom) score 3.

Study Setting. 47 VA Medical Centers will recruit on average 100 patients/site over 3 years. These recruitment sites, which have already been identified, have adequate numbers of cirrhosis patients eligible for screening, a qualified hepatologist and radiologist to serve as local site investigators (LSIs), adequate MRI and US capacity, and access to a multidisciplinary liver tumor board (MLTB).

Target Sample Size. N=2350 per group, total N=4700.

Randomization. The randomization scheme will be random permuted with variable block size and will be stratified by medical center and MELD score.

Intervention. Participants will be randomized in a 1:1 ratio to one of two screening arms:

a. Abdominal aMRI+ serum AFP every 6 months, OR b. Abdominal US+ serum AFP every 6 months, from the time of recruitment until the end of study Year 8.

The aMRI protocol will include only T1-weighted pre-contrast and dynamic contrast-enhanced images utilizing an extracellular gadolinium-based contrast agent. aMRI takes only ~15 minutes to perform. Enrollment will occur in Years 1-3, screening per protocol will continue through Year 8, and follow-up for mortality will continue through Year 8. Analysis and publication will be in Year 9.

Primary Outcome. HCC-related mortality.

Power Calculations. The study is powered to detect a minimum relative reduction in HCC-related mortality of 35% in the aMRI+AFP arm compared to the US+AFP arm, i.e. a reduction in cumulative HCC-related mortality at Year 8 from 7.1 per 100 patients in the US+AFP arm to 4.6 per 100 patients in the aMRI+AFP arm (absolute difference in HCC-related mortality of 2.5 per 100 patients), adjusted for dropout due to death from other causes or withdrawals, with power 88% and two-sided alpha 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Cirrhosis due to any underlying etiology diagnosed by one or more of the following:

   * Histology of liver biopsy
   * Radiologic criteria (nodular liver, evidence of portal hypertension)
   * Clinical signs of cirrhosis (gastroesophageal varices, ascites, hepatic encephalopathy)
   * Vibration controlled transient elastography (VCTE, specifically Fibroscan, which is available in all participating sites) with liver stiffness >12.5kPa or magnetic resonance elastography >5.0 kPa
2. High Risk of Liver Cancer: This will be defined by one or more of the following:

   * Current HCV infection (detectable HCV RNA)
   * FIB-4 score 3.25, within 6 months of randomization
   * Estimated annual HCC incidence >2.5%, within 6 months of randomization, calculated by VA-specific models that the investigators developed (available on the national VA ALD Dashboard and at www.hccrisk.com).
3. Age 18-75
4. Able to provide informed consent

Exclusion Criteria:

1. Prior diagnosis or of HCC
2. Current suspicion of HCC
3. Prior receipt of organ transplantation
4. Currently listed for organ transplantation.
5. Participation in a conflicting HCC screening trial
6. Advanced liver dysfunction, defined by Child C Cirrhosis (CTP score 10), or MELD score >20, within 6 months prior to randomization
7. Glomerular Filtration Rate (GFR) <30 ml/min
8. Multiple comorbid conditions resulting in limited life expectancy, defined by a cirrhosis-specific comorbidity index (CirCom)112 score 3. Of note, early stage malignancies of the bladder, lung, or prostate will not be excluded.
9. Estimated life expectancy <5 years as determined by the clinical judgement of the Study Investigator
10. Contraindications to undergoing contrast-enhanced MRI:

    * Allergy to gadolinium-based contrast agents
    * MRI-incompatible implantable devices (e.g. pacemakers, defibrillators, resynchronization devices)
    * Implantable neurostimulation device
    * Implantable cochlear implant/ear implant
    * Drug infusion pumps (e.g. insulin pump, analgesic or chemotherapy pumps)
    * Metallic foreign bodies in or around the eye
    * Metallic fragments, such as bullets, shotgun pellets or shrapnel
    * Metallic body piercings that cannot be removed
    * Cerebral artery aneurysm clips
    * Severe claustrophobia
    * Unable to fit on MRI machine due to weight (weight >400lbs) or body habitus
11. Inability to complete planned study visits (e.g. lives too far from VA, no transportation, etc.)
12. Currently pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4700 (Estimated)
Dates: Start 2023-11-03 (Actual); Primary Completion 2030-09-01 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
Hepatocellular Carcinoma Mortality | 8 years
  death due to liver cancer

SECONDARY OUTCOMES:
Stage of Hepatocellular Carcinoma at diagnosis | 8 years
  Stage of Hepatocellular Carcinoma at time of diagnosis
Receipt of potentially curative treatments for Hepatocellular Carcinoma | 8 years
  Receipt of potentially curative treatments for Hepatocellular Carcinoma
Overall Survival | 8 years
  overall survival of liver cancer

CONTACTS AND LOCATIONS:
Overall Officials: George N. Ioannou, MD MS, Study Chair — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (17):
- United States (17):
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA Northern California Health Care System, Mather, CA, Sacramento, California
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE, Omaha, Nebraska
  - James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington
  - William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ioannou GN, Taddei TH, Planeta BM, Huang GD, Weiss NS, Morgan TR, Dominitz JA, Abou-Alfa GK, Bashir MR, Beheshti MV, Singal AG, Moylan CA, Boland RJ, Buchwalder LF, Mehta RL, Hoisington KS, Do NV, Rogal SS, Kaplan DE, Benhammou JN, Su GL, McDonald LM, Dani G, Dunn DP, Chang ST, Onyiuke IY, Sharma A, Kyriakides TC; PREMIUM Study Group. Practice changing RCT design and rationale: Abbreviated MRI plus AFP vs. ultrasound plus AFP for HCC surveillance in cirrhosis (PREMIUM study). JHEP Rep. 2025 Nov 6;8(2):101666. doi: 10.1016/j.jhepr.2025.101666. eCollection 2026 Feb. PMID 41624484